CLINICAL TRIAL: NCT01765244
Title: Multicenter Clinical Trial to Evaluate the Safety and Feasibility of an Allogeneic Tissue Engineered Drug (Nanostructured Artificial Human Cornea) in Patients With Corneal Trophic Ulcers Refractory to Conventional Treatment
Brief Title: Allogeneic Tissue Engineering (Nanostructured Artificial Human Cornea) in Patients With Corneal Trophic Ulcers in Advanced Stages, Refractory to Conventional (Ophthalmic) Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAH/Ulc/2010; 2010-024290-40 (EudraCT Number)
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Severe Trophic Corneal Ulcers Refractory to Conventional Treatment; Sequelae of Previous Trophic Corneal Ulcers
Keywords: Corneal trophic ulcers, limbal deficiency, cornea blindness

STUDY DESIGN:
Intervention Model Description: Bioengineered anterior human corneal substitute Amniotic membrane corneal graft
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior lamellar nanostructured artificial human cornea (Experimental): Anterior lamellar nanostructured artificial human cornea with allogenic from dead donor and cultured in its inside and allogeneic corneal epithelium cultured in its surface
  Interventions: Drug: Anterior lamellar nanostructured artificial human cornea.
- Amniotic membrane transplantation (Active Comparator): Amniotic membrane transplantation as conventional treatment of corneal trophic ulcers.
  Interventions: Other: Amniotic membrane transplantation

INTERVENTIONS:
Drug: Anterior lamellar nanostructured artificial human cornea. — Implantation of an anterior lamellar nanostructured artificial human cornea with allogeneic cells from dead donors embedded in a fibrin-agarose scaffold
  Other Names: Bioengineered human anterior corneal substitute
  Arms: Anterior lamellar nanostructured artificial human cornea
Other: Amniotic membrane transplantation — Implantation of an amniotic membrane graft to cover the corneal scarring using the mixed graft/patch technique.
  Arms: Amniotic membrane transplantation

SUMMARY:
This is a prospective, phase I-II, randomised, open-label clinical trial that will evaluate the safety and feasibility, as well as clinical efficacy evidence, of a bioengineered anterior corneal substitute in adults with severe trophic corneal ulcers. This model of human anterior allogeneic cornea will provide an alternative approach in cases where human donor keratoplasty is not an option.

DETAILED DESCRIPTION:
This is a phase I-II, randomised, controlled, open-label clinical trial, currently ongoing in eleven Spanish hospitals, to evaluate the safety and feasibility, as well as clinical efficacy evidence, of a bioengineered human anterior corneal substitute in adults with severe trophic corneal ulcers refractory to conventional treatment, or with sequelae of previous ulcers. In the initial phase of the trial (n=5), patients were sequentially recruited, with a safety period of 45 days, receiving the bioengineered corneal graft. In the second phase of the trial (currently ongoing), subjects are block randomised (2:1) to receive either the corneal graft (n=10), or amniotic membrane (n=5), as the control treatment. Adverse events, implant status, infection signs and induced neovascularization are evaluated as determinants of safety and feasibility of the bioengineered graft (main outcomes). Study endpoints are measured along a follow-up period of 24 months, including 27 post-implant assessment visits according to a decreasing frequency. Intention to treat, and per protocol, and safety analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged≥18, with no upper age limit.
* Patients that give their informed consent for study participation.
* Stage 3 Mackie corneal ulcers that do not respond to conventional medical treatment, or patients having undergone previous stage 3 Mackie corneal ulcers,33 currently suffering sequelae such as stromal fibrosis or corneal thinning, having no effective therapeutic alternative.
* Stromal involvement, not reaching the Descemet membrane. Central or peripheral localization.
* Minimum duration of the disease causing the corneal ulcer: 6 weeks.
* No active ocular infection.
* Patients with normal laboratory parameters as defined by: Leukocytes≥3000 cells/µL; Neutrophils≥1500 cells/µL; Platelets≥100 billion/L; AST/ALT≤1.5 ULN; Creatinine≤1.5 mg/dL.

Exclusion Criteria:

* Absence of stromal involvement.
* Good response to standard medical treatments for corneal disease in less than 3 to 5 weeks.
* Bullous keratopathy or other endothelial decompensations.
* Active ocular infection.
* Positive serology to HBV, HCV, HIV or any other pathology that may interfere with correct patient follow-up.
* Pregnant or breast-feeding women or childbearing-age women that do not consent the use of contraceptive methods approved in the protocol.
* Medical history of active neoplasia within the past 5 years. Participation in other clinical trials in 3 months previous to inclusion, or in the previous 5 years for trials with advanced therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01-17 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Adverse events (and serious adverse events) causally related to experimental treatment. | 24 months
Implant status (integrity, detachment and reabsorption) | 24 months
Local, regional or systemic infections related with the implant | 24 months
Induced corneal neovascularization | 24 months

SECONDARY OUTCOMES:
Ulcer persistency or relapse and corneal stromal repair | 24 months
Visual acuity | 24 months
Corneal transparency | 24 months
Tear function (TBUT and Schirmer) | 24 months
Quality of life (EQ-5) | 24 months
Induced chronic ocular complications | 24 months
In vivo confocal microscopy (IVCM) analysis of the grafted bioengineered cornea (and AM) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Medialdea, MD, PhD, Study Director — Hospital U Virgen de las Nieves; Miguel Alaminos, MD, PhD, Study Chair — Universidad de Granada
Locations (11):
- Spain (11):
  - Hospital San Juan de Dios, Bormujos
  - University Hospital Puerta del Mar, Cadiz
  - Hospital la Arruzafa, Córdoba
  - Hospital Universitario Reina Sofía, Córdoba
  - University Hospital San Cecilio, Granada
  - University Hospital Virgen de las Nieves, Granada
  - Hospital Costa del Sol, Marbella
  - Marina Rodriguez Calvo-Mora, Málaga
  - University Hospital Virgen Macarena, Seville
  - University Hospital Virgen de Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville

REFERENCES:
- [Background] Gonzalez-Andrades M, Mata R, Gonzalez-Gallardo MDC, Medialdea S, Arias-Santiago S, Martinez-Atienza J, Ruiz-Garcia A, Perez-Fajardo L, Lizana-Moreno A, Garzon I, Campos A, Alaminos M, Carmona G, Cuende N. A study protocol for a multicentre randomised clinical trial evaluating the safety and feasibility of a bioengineered human allogeneic nanostructured anterior cornea in patients with advanced corneal trophic ulcers refractory to conventional treatment. BMJ Open. 2017 Sep 24;7(9):e016487. doi: 10.1136/bmjopen-2017-016487. PMID 28947445